CLINICAL TRIAL: NCT03495349
Title: Effectiveness and Safety of Antibiotherapy in Diabetic Patients Treated for a Diabetic Foot Infection.
Acronym: DIABASE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0850
Record Dates: First submitted 2018-03-12; First posted 2018-04-12 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Foot Infection
MeSH Terms: interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic foot infection: All of the patients followed for a diabetic foot infection in Hospices Civils of Lyon
  Interventions: Other: safety and effectiveness of the usual treatments of diabetic foot infections

INTERVENTIONS:
Other: safety and effectiveness of the usual treatments of diabetic foot infections — clinical and biological follow-up necessary to assess the safety and effectiveness of the medical treatments, MOS-SF survey (36-Item Short Form Survey) to study the quality of life.

SUMMARY:
Diabetes is a frequent and serious disease, with many complications. Diabetic foot ulcers are a frequent complication. Infection of diabetic foot ulcers is common, and requires heavy medical and/or surgical treatments. Antibiotherapy is one of the main options for the treatment of the diabetic foot ulcers, but it has many side effects.

The aim of this study is to evaluate effectiveness and safety of medical treatments, in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults men and women
* Followed for diabetic foot infection (grades 2 to 4 of IWGDF classification)
* That accepted to take part in the study

Exclusion Criteria:

* Legal safeguard
* Pregnant women
* Patient that can't accept to take part in the study because can't be informed
* Exclusive surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the patients followed and treated for diabetic foot infection in the 2 Endocrinology departments of Hospices Civils of Lyon. All of the patients have accepted to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of adverse effects in patients treated by antibiotherapy for diabetic foot infection, assessed by clinical or biological methods | 1 year
  Effectiveness :
  * For soft tissue infections, remission is defined by the disappearance of any functional or physical sign of infection,
  * For osteomyelitis, remission is defined as the absence of clinical and /or radiological recurrence at the initial site one year after antibiotic therapy cessation.
Occurrence of adverse effects in patients treated by antibiotherapy for diabetic foot infection, assessed by clinical or biological methods | 1 year
  Occurrence of side effects:
  All clinical and/or biological adverse events will be reported. The severity of any adverse events will be graded according to the criteria of Common Terminology Criteria for Adverse Events (CTCAE) from grade 1 (mild) to 5 (death).
  Clinical adverse events included gastrointestinal disorders, skin eruption, pain, weight gain or loss Biological adverse events included impair kidney function, increase liver serum markers, anemia, low neutrophils count, thrombopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Vouillarmet, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Groupement Hospitalier Est, Bron
  - Centre Hospitalier Lyon Sud, Pierre-Bénite